CLINICAL TRIAL: NCT02997111
Title: Is the PFA-100 Responsive to the Effect of Energy Drinks on Platelet Function Changes?
Brief Title: PFA-100 Responsive to Effect of Energy Drinks on Platelet Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Katherine Newsham PhD, ATC, Associate Professor, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 27619
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Platelet Function; Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Energy drink (Other): Single group study. Platelet function analyzed with PFA-100 before and 60 minutes after ingestion of 250 ml sugar-free energy drink
  Interventions: Device: PFA-100

INTERVENTIONS:
Device: PFA-100 — The PFA-100 will be used to assess platelet function before and after energy drink consumption.
  Other Names: Platelet function analyzer

SUMMARY:
This study evaluates the responsiveness of the Platelet Function Analyzer (PFA-100) to the effect of energy drinks on platelet function. Participants' will have blood drawn prior to and 60 minutes after ingesting 250ml of a commercially available sugar-free energy drink.

DETAILED DESCRIPTION:
Two previous studies have demonstrated increased platelet aggregation 60 minutes after drinking a commercially available sugar-free energy drink. These studies utilized traditional platelet function studies, such as light transmission aggregometry (LTA), where platelet function is examined while adding varying concentrations of a panel of agonist to platelets. These studies are technically difficult, time intensive studies requiring specialized laboratories. They are relatively non-physiologic and do not mimic platelet response to vessel wall damage. Other tests better represent the reactions to vessel wall damage, including the PFA-100, which measures platelet aggregation and adhesion under conditions of high shear.

Overall, PFA-100 is less expensive, requires less technical skill, and is less time consuming than LTA. It has been utilized in bleeding disorders and is demonstrating promise as a marker of thrombophilia. PFA-100 has demonstrated sensitivity to drug and dietary effects. It has also shown differences in closure time between sedentary and athletic individuals PFA-100 has not been used to investigate the effect of energy drinks.

ELIGIBILITY:
Inclusion Criteria:

* a history of consuming at least one energy drink beverage in the past 6 months without adverse effects;
* engage in moderate to strenuous physical activity more than 3 days per week.

Exclusion Criteria:

* Known thromboembolic risk including protein C or S deficiency, anti-thrombin III deficiency, Factor V Leiden;
* history of thromboembolic event;
* current or previous anti-coagulation therapy, anti-platelet therapy, calcium antagonists; - current tricyclic antidepressant therapy, current selective serotonin re-uptake inhibitor therapy; antibiotic therapy; or famotidine therapy;
* acute illness;
* pregnancy;
* hemophilia;
* significant history of cardiovascular disease and/or diabetes mellitus;
* history of adverse effect of energy drinks.
* Inability to comply with pre-test dietary and activity requirements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Closure time | one hour
  Agonist induced platelet activation and aggregation resulting in occlusion of the aperture and cessation of blood flow termed the closure time

SECONDARY OUTCOMES:
blood pressure | one hour (every 15 minutes)
pulse | one hour (every 15 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Newsham, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data with other researchers